CLINICAL TRIAL: NCT00005845
Title: Phase I Study of the Farnesyl Transferase Inhibitor R115777 (NSC #702818) in Patients With Myelodysplastic Syndrome
Brief Title: Tipifarnib in Treating Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01158; NCI-2009-01158 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000067862; DM01-582 (Other: M D Anderson Cancer Center); 5625 (Other: CTEP); U01CA062461 (NIH)
Record Dates: First submitted 2000-06-02; First posted 2003-08-29 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Myelomonocytic Leukemia; de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Refractory Anemia; Refractory Anemia With Excess Blasts; Refractory Anemia With Excess Blasts in Transformation; Refractory Anemia With Ringed Sideroblasts; Refractory Cytopenia With Multilineage Dysplasia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Anemia, Refractory; Anemia, Refractory, with Excess of Blasts | interventions — tipifarnib

ARMS (1):
- Treatment (tipifarnib) (Experimental): Patients receive tipifarnib PO BID on weeks 1, 3, 5, and 7. Treatment repeats every 8 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tipifarnib; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: tipifarnib — Given PO
  Other Names: R115777; Zarnestra
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial studies the side effects and best dose of tipifarnib in treating patients with myelodysplastic syndromes. Tipifarnib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicity profile and antitumor activity of the farnesyltransferase (FTase) inhibitor R115777 (tipifarnib) in patients with myelodysplastic syndrome (MDS) treated on a one week on/one week off schedule.

II. To determine the effect on R115777 on a one week on/one week off schedule on FTase activity, prenylation of RAS and other substrates and on downstream effects.

OUTLINE: This is a dose-escalation study.

Patients receive tipifarnib orally (PO) twice daily (BID) on weeks 1, 3, 5, and 7. Treatment repeats every 8 weeks for up to 2 courses in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically MDS (including French-American-British [FAB] types refractory anemia [RA], refractory anemia with ringed sideroblasts [RARS], refractory anemia with excess blasts [RAEB], refractory anemia with excess blasts in transformation [RAEBT], or chronic myelomonocytic leukemia [CMMoL]); for the purpose of the study, all patients will be classified by World Health Organization (WHO) criteria

  * By these criteria, FAB RA are split into:
  * Pure dyserythropoietic refractory anemia (PRA)

    * Refractory cytopenia with multilineage dysplasia (RCMD)
  * FAB RARS is split into:

    * Pure sideroblastic anemia (PSA)
    * Refractory sideroblastic cytopenia with multilineage dysplasia (RSCMD)
  * FAB RAEB is split into:

    * RAEB I (< 10% BM blasts)
    * RAEB II (10-20% BM blasts)
  * Patients with CMMoL, and RAEBT by FAB classification will be included in the protocol
* Prognosis will be assessed by International Prognostic Scoring System (IPSS) criteria
* =< 2 prior therapies
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Life expectancy of greater than 12 weeks
* Bilirubin =< 1.5mg %
* Creatinine =< 1.5mg %
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (3 months for UCN01) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to R115777 (such as imidazoles)
* Patients eligible for bone marrow transplant (=< 60 years old), with a compatible sibling, no contraindications for transplant
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with R115777.
* Growth factors other than filgrastim (G-CSF) are excluded; patients should be off excluded growth factors for 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2002-06; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
MTD defined as the next lower dose level at which 2 patients experience dose limiting toxicity (DLT) defined as grade 3 or 4 toxicity according to the Cancer Therapy Evaluation Program Common Toxicity Criteria | Up to 8.5 years
  The final analysis will report all toxicities by grade, dose, cycle, and by cumulative dose.
Response rate | Up to 8.5 years
  Will be reported overall and by dose level.

SECONDARY OUTCOMES:
FTase inhibition | Up to 8.5 years
  Based on the shape of the relationship (e.g. linear vs saturation vs peak), a dose response analysis will be performed to describe/summarize the relationship (correlation analysis or curve-fitting).
Accumulation of unfarnesylated lamin B1 | Up to 8.5 years
  Based on the shape of the relationship (e.g. linear vs saturation vs peak), a dose response analysis will be performed to describe/summarize the relationship (correlation analysis or curve-fitting).
Accumulation of RAS proteins | Up to 8.5 years
  Based on the shape of the relationship (e.g. linear vs saturation vs peak), a dose response analysis will be performed to describe/summarize the relationship (correlation analysis or curve-fitting).

CONTACTS AND LOCATIONS:
Overall Officials: Razelle Kurzrock, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States